CLINICAL TRIAL: NCT00224549
Title: Management of Resistant Hypertension -Pharmacokinetic Assessment of Different Antihypertensive Regimen -Comparison of Two Treatment Strategies: Increase Sodium Depletion or Combined Blockage of Renin-angiotensin System (RAS)
Brief Title: PHARES Study: Management of Resistant Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040407
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2007-03

CONDITIONS: Hypertension
Keywords: Resistant hypertension; Combined diuretic therapy; Combined RAS blockers
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irbesartan, amlodipine and hydrochlorothiazide — irbesartan, amlodipine and hydrochlorothiazide

SUMMARY:
The purpose of this study is to assess the efficacy of two different treatment regimens for treating resistant hypertension previously uncontrolled with at least 3 antihypertensive treatments. The study hypothesis is that these two regimens (one based on increasing diuretics and the other based on increasing renin angiotensin system blockage) may not differ in terms of efficacy.

DETAILED DESCRIPTION:
Tested hypothesis: For essential resistant hypertension, a new regimen based on intensive RAS blockage is non inferior to the recommended regimen based on intensive sodium depletion.

Primary objective: To demonstrate non-inferiority (i.e difference between the two regimen less than 5 mmHg for the mean day-time SBP at week 12)

* One treatment arm including irbesartan 300 mg, hydrochlorothiazide (HCTZ) 12.5mg, amlodipine 5 mg, ramipril 10mg and bisoprolol 10 mg
* One treatment arm including irbesartan 300 mg, HCTZ 12.5mg, amlodipine 5 mg, spironolactone 25 mg, furosemide 40 mg and amiloride 5 mg.

Secondary objectives:

* To assess clinical and biological safety and efficacy of these regimen
* To evaluate predicted factors of controlled or uncontrolled BP
* To evaluate compliance to treatment
* To compare the cost of the different strategies
* To compare the two strategies in terms of endothelial function and left ventricular diastolic filling

Study design:

* Period 1 from week-4 to week 0 : 4-week treatment for all patients with irbesartan 300 mg, HCTZ 12.5mg, amlodipine 5 mg. At the end of this period, an ABPM will be performed: only patients with a mean day time SBP>135 and/or DBP>85 mmHg will be randomized for a further 3 months treatment
* Period 2 from week 0 to week 4: patients will be randomized in two groups, the first one receiving spironolactone 25mg and the second one receiving ramipril 5 mg as add-on therapy (on top of the previous tri-therapy).
* Period 3 from week 4 to week 8: Patients with BP controlled at week 4 (i.e mean home blood pressure measurement (HBPM) <135/85 mmHg at week 4) remain on the same treatment. For those uncontrolled (i.e. mean HBPM >135/85 mmHg at week 4), furosemide 20 mg will be added in the first group and ramipril will be titrated to 10 mg in the second group
* Period 4 from week 8 to week 10: Patients with BP controlled at week 8 (i.e. mean HBPM <135/85 mmHg at week 8) remain on the same treatment. For those uncontrolled (i.e. mean HBPM >135/85 mmHg at week 8), furosemide will be titrated to 40 mg in the first group and bisoprolol 5 mg will be added in the second group.
* Period 5 from week 10 to week 12 (end of the study): Patients with BP controlled at week 10 (i.e mean HBPM <135/85 mmHg at week 10) remain on the same treatment. For those uncontrolled (i.e mean HBPM > 135/85 mmHg at week 10), amiloride 5 mg will be added to the previous treatment in the first group and bisoprolol will be titrated to 10 mg in the second group.

Reasons for treatment discontinuation:

* Patient decision
* Informed consent withdrawal
* SBP>180 mmHg or <100 mmHg (HBPM) whatever the time during the trial
* Adverse events related to treatment or not

ELIGIBILITY:
Inclusion Criteria:

* Primary hypertension
* Resistant hypertension defined by mean day-time SBP > 135 mmHg and DBP > 85 mmHg (determined with ABPM device) after a standardized 4-week regimen including irbesartan, amlodipine and HCTZ.

Exclusion Criteria:

* Secondary hypertension
* Unstable angina, history of stroke or coronary heart disease (coronary by-pass or angioplasty) in the previous 3 months
* History of cough with ACEi or gynecomastia with antialdosterones
* Heart failure (New York Heart Association [NYHA] III-IV)
* Contraindication to beta blockers because of bronchopathy or auriculoventricular block
* Diabetes mellitus (type 1 or 2) with HbA1C > 8%
* Renal failure with creatinine clearance < 40ml/min (COCKROFT evaluation)
* Arm circumference > 42 cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Mean day-time systolic blood pressure (SBP) at week 12, measured with an average blood pressure measurement (ABPM) device | at week 12
  Mean day-time systolic blood pressure (SBP) at week 12, measured with an average blood pressure measurement (ABPM) device

SECONDARY OUTCOMES:
Efficacy: mean day-time diastolic blood pressure (DBP) at week 12, mean 24 hours SBP and DBP at week 12 measured with an ABPM device | at week 12,
  hours SBP and DBP at week 12 measured with an ABPM device
Safety and tolerability: | during the study
  Safety and tolerability:
During the study BP will be evaluated every 4 weeks by home blood pressure measurement [HBPM] in order to detect hypotension) | every 4 weeks
  During the study BP will be evaluated every 4 weeks by home blood pressure measurement [HBPM] in order to detect hypotension)
Biological examinations: | during the study
  Biological examinations:
blood and urinary electrolytes with creatinemia at week 0, 4, 8, 10 and 12 | at week 0, 4, 8, 10 and 12
  blood and urinary electrolytes with creatinemia at week 0, 4, 8, 10 and 12
brain natriuretic peptide (BNP), active renin, aldosterone at week 0 and 12 | at week 0 and 12
  brain natriuretic peptide (BNP), active renin, aldosterone at week 0 and 12
Other explorations: | during
  Other explorations:
Treatment compliance (study drug accounting, N-acetyl-seryl-aspartyl-lysyl-proline [Ac SDKP] for angiotensin converting enzyme inhibitor [ACEi]) | during the study
  Treatment compliance (study drug accounting, N-acetyl-seryl-aspartyl-lysyl-proline [Ac SDKP] for angiotensin converting enzyme inhibitor [ACEi])
Echocardiography (week 0 and 12) | week 0 and 12
  Echocardiography (week 0 and 12)
Endothelial function (week 0 and 12) | week 0 and 12
  Endothelial function (week 0 and 12)
Pharmacokinetics of drugs (week 0 and 12) | week 0 and 12
  Pharmacokinetics of drugs (week 0 and 12)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOBRIE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Investigation Clinical Center European Georges Pompidou Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Mendes M, Dubourg J, Blanchard A, Bergerot D, Courand PY, Forni V, Frank M, Bobrie G, Menard J, Azizi M. Copeptin is increased in resistant hypertension. J Hypertens. 2016 Dec;34(12):2458-2464. doi: 10.1097/HJH.0000000000001106. PMID 27755389
- [Derived] Frank M, Peyrard S, Bobrie G, Azizi M. Method of mean value calculation as an additional source of variability in ambulatory blood pressure measurement. Am J Hypertens. 2010 Jul;23(7):725-31. doi: 10.1038/ajh.2010.47. Epub 2010 Mar 25. PMID 20339354